CLINICAL TRIAL: NCT04913389
Title: Novel Approach to Prevention of Altitude-related Illness in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Acetazolamide to Prevent Impending Altitude-illness in Patients With COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine, Kyrgyz Republic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01-2021-KEB
Record Dates: First submitted 2021-05-23; First posted 2021-06-04 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Altitude Sickness; Altitude Hypoxia
Keywords: Acetazolamide; Mountain sickness; Hypoxemia; Prevention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Altitude Sickness; Hypoxia | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent pharmacist will prepare identically looking active and placebo capsules labelled with secret codes. Codes will be concealed to investigators and patients until completion of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetazolamide (Active Comparator): Acetazolamide (oral capsules)
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo (oral capsules)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide (oral capsules @125 mg), starting dose 3 capsules (375 mg), subsequent doses 1 capsule (125 mg) in the morning, 2 capsules (250 mg) in the evening, administered in qualifying participants, during the stay at 3100 m.
  Other Names: Acetazolamide, oral capsule
  Arms: Acetazolamide
Drug: Placebo — Placebo (oral capsules, identically looking as active drug), starting dose 3 capsules, subsequent doses 1 capsule in the morning, 2 capsules in the evening, administered in qualifying participants, during the stay at 3100 m.
  Other Names: Placebo, oral capsule
  Arms: Placebo

SUMMARY:
The purpose of this randomized, placebo-controlled double-blind trial is to evaluate efficacy of acetazolamide in preventing overt altitude-related adverse health effects (ARAHE) in lowlanders with chronic obstructive pulmonary disease (COPD) developing early signs of altitude-illness during altitude travel.

DETAILED DESCRIPTION:
This randomized placebo-controlled, double-blind, parallel-design trial will evaluate effectiveness of acetazolamide in reducing the incidence of predefined altitude-related adverse health effects in lowlanders with chronic obstructive pulmonary disease (COPD) travelling to high altitude and developping early symptoms and/or signs of impending altitude-illness. Qualifying participants will be randomized 1:1 to acetazolamide or placebo treatment during their further stay of 2 days at 3'100 m.

An interim-analysis will be performed after the first year of the study or when 38 participants are randomized, whichever comes first. Symmetric stopping boundaries at P<0.001 will be applied (Peto approach).

ELIGIBILITY:
Inclusion criteria

* Men and women, age 35-75 y, living at low altitude (<800 m).
* COPD diagnosed according to the Global Initiative for Obstructive Lung Disease (GOLD) guidelines, forced expiratory volume in one second 40-80% predicted, pulse oximetry ≥92%, PaCO2 <6 kilopascal, breathing ambient air at 760 m.
* One of the following early signs and/or symptoms of impending altitude-illness identified by self-monitoring during ascent to or stay at 3100 m:

  * Pulse oximetry SpO2≤84%
  * Headache or nausea/vomiting or fatigue/weakness or dizziness/light-headedness of at least moderate intensity

Exclusion criteria

* COPD exacerbation, very severe COPD with hypoxemia or hypercapnia at 760 m (see above).
* Other lung disease, relevant comorbidities (such as uncontrolled cardiovascular disease, i.e., unstable arterial hypertension, coronary artery disease; previous stroke; obesity (body mass index >35 kg/m2); internal, neurologic, rheumatologic or psychiatric disease; current heavy smoking (>20 cigarettes per day).
* Renal failure and/or allergy to sulfonamides.
* Patients who do not have early signs and/or signs of impending altitude-illness by self-monitoring (as defined above) at 3'100m will not be included.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of altitude-related adverse health effects | Day 1 to 3 at 3'100m
  Difference between participants receiving acetazolamide and placebo in the incidence of altitude-related adverse health effects defined as:
  * Moderate to severe acute mountain sickness (Lake Louise score >4 including headache and/or Acute Mountain Sickness cerebral score ≥0.7)
  * Severe hypoxemia (SpO2 at rest <80% for >30 min; or SpO2 <75% for >15 min; or exercise oxygen desaturation SpO2 <75% for >1 min accompanied by symptoms or signs of hypoxemia)
  * Symptomatic cardiovascular disease (arterial blood pressure systolic >200 mmHg, diastolic >120 mmHg, chest pain with ECG signs of cardiac ischemia)
  * New onset neurologic impairment
  * Other intercurrent illness requiring medical treatment
  * Any discomfort leading to the wish of a patient to return to low altitude or withdraw from the study by the independent physician

SECONDARY OUTCOMES:
Incidence and severity of the individual components of altitude-related adverse health effects | Day 1 to 3 at 3'100m
  Difference between participants receiving acetazolamide and placebo in the incidence and severity of components of altitude-related adverse health effects
Arterial blood gases | Day 2 at 3'100 m
  Difference between participants receiving acetazolamide and placebo in arterial blood gases
Forced expiratory volume in one second (FEV1) | Day 2 at 3'100 m
  Difference between participants receiving acetazolamide and placebo in forced expiratory volume in one second (FEV1) measured by spirometry
Forced vital capacity (FVC) | Day 2 at 3'100 m
  Difference between participants receiving acetazolamide and placebo in forced vital capacity (FVC) measured by spirometry
Drug side effects | Day 1 to 3 at 3'100m
  Difference between participants receiving acetazolamide and placebo in the incidence of drug side effects

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, Study Chair — University Hospital, Zürich, Switzerland; Talant M Sooronbaev, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan; Michael Furian, Principal Investigator — University Hospital, Zürich
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan